CLINICAL TRIAL: NCT00794989
Title: A Study Evaluating the Effect of Flaxseed on Biomarkers of Breast Cancer Risk
Brief Title: Flaxseed in Preventing Breast Cancer in Premenopausal Women at Risk of Developing Breast Cancer
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: low accrual
Sponsor: Roswell Park Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: I 81906; RPCI-I-81906 (Other: Roswell Park Cancer Institute); 11-0575 (Other: University of Chicago)
Record Dates: First submitted 2008-11-20; First posted 2008-11-21 (Estimated); Last update posted 2016-06-03 (Estimated); Status verified 2016-06

CONDITIONS: Breast Cancer; Precancerous Condition
Keywords: breast cancer; atypical ductal breast hyperplasia; lobular breast carcinoma in situ; ductal breast carcinoma in situ; breast cancer prevention; high risk breast cancer
MeSH Terms: conditions — Breast Neoplasms; Precancerous Conditions; Carcinoma, Intraductal, Noninfiltrating; Breast Carcinoma In Situ

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm 1: Intervention (Experimental): Patients ingest ground flaxseed daily, with already prepared foods, for 6 months.
  Interventions: Dietary Supplement: Ground Flaxseed
- Arm 2: Observational (Other): Patients do not receive ground flaxseed.
  Interventions: Other: No Intervention

INTERVENTIONS:
Dietary Supplement: Ground Flaxseed — Given orally
  Arms: Arm 1: Intervention
Other: No Intervention — Participants randomized to Arm 2 do not receive any intervention
  Arms: Arm 2: Observational

SUMMARY:
RATIONALE: Ground flaxseed may prevent breast cancer in premenopausal women at increased risk of developing primary breast cancer.

PURPOSE: This randomized clinical trial is studying how well flaxseed works in preventing breast cancer in premenopausal women at risk of breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary aims:

* Determine if 25 grams of flaxseed supplementation daily

  * modifies proliferation (ki-67) and apoptotic rates after six months
  * modifies expression of estrogen regulated genes: Cyclin D1, survivin, and VEGF at six months
  * modifies serum IGF-1 and serum binding protein (IGFBP)-3 levels from baseline to 6 months
  * and evaluate the feasibility and tolerability of flaxseed consumption, and determine factors that lead to decreased compliance

STUDY OUTLINE:

This is a randomized study. Patients are randomized to 1 of 2 arms.

* Arm I (intervention): Patients ingest 25 grams ground flaxseed daily, with already prepared foods, for 6 months. Patients are instructed to record the time and with what foods flaxseed is consumed, and the number of bowel movements daily. Throughout the 6-month intervention period, patients also complete unannounced telephone-administered surveys recounting all foods and beverages consumed within the previous 24 hours.
* Arm II (observation): Patients do not receive ground flaxseed. All patients complete a diary about menstrual cycle duration and presence or improvement of premenstrual symptoms (e.g., cramping, bloating, headache, insomnia, or other irregular symptoms). Patients also complete questionnaires at 1, 3, and 6 months to access changes in diet, physical activity, menstrual history, demographic characteristics, and medical history and a specimen questionnaire at baseline and at 1, 3, and 6 months.

Blood and first-void urine samples are collected at baseline and at 1, 3, and 6 months to measure levels of lignan metabolites, flaxseed compliance, serum thiocyanate, malondialdehyde, and for biomarker studies by capillary gas chromatography-mass spectrometry, high-performance liquid chromatography, and ELISA.

After completion of study therapy, patients are followed monthly for up to 6 months.

ELIGIBILITY:
* Patients enrolled in must meet ≥ 1 of the following criteria:

  * History of unilateral or bilateral atypical ductal hyperplasia with or without family history
  * History of atypical lobular hyperplasia or lobular carcinoma in situ with or without family history
  * History of ductal carcinoma in situ
  * Prior stage I breast cancer allowed provided it was adequately treated and therapy was completed ≥ 1 year ago
  * Lifetime risk for developing breast cancer > 20% (based on Gail or Claus model)
  * No abnormal mammogram requiring short-term follow-up within the past 6 months
  * No severe atypia or carcinoma cells on RPRNA

PATIENT CHARACTERISTICS:

* Premenopausal
* ECOG performance status 0-1
* Patients enrolled must meet the following criteria:

  * No peri- or postmenopausal status as determined by estradiol levels < 20 ng/dL and FSH levels > 45 ng/dL
  * No thrombocytopenia (defined as platelet count < 50,000/mm^3)
  * Creatinine ≤ 1.5 mg/dL
  * Not pregnant or nursing
  * Fertile patients must use effective contraception consistently
  * No other prior malignancy allowed except for the following:

    * Basal cell or squamous cell carcinoma
    * In situ cervical cancer
  * No history of any of the following conditions within the past 5 years:

    * Crohn disease
    * Ulcerative colitis
    * Inflammatory bowel disease
    * Irritable bowel syndrome
    * Celiac sprue
    * Malabsorption syndrome
    * Diverticulitis
    * Diverticulosis
  * No allergy to flaxseed, other seeds or nuts, or wheat

PRIOR CONCURRENT THERAPY:

* Patients enrolled in part 1 must meet the following criteria:

  * No prior breast implants or tram-flap reconstruction

    * Breast reduction allowed
  * No prior neoadjuvant chemotherapy or other chemotherapy within the past year
  * No prior neoadjuvant hormonal therapy
  * No prior whole radiation to the contralateral breast undergoing random periareolar fine needle aspiration (RPFNA)
  * No concurrent coumadin or other chronic anticoagulants (even if they are held for surgery)
* Patients enrolled in part 2 must meet the following criteria:

  * More than 1 year since prior chemotherapy and adjuvant hormonal therapy for breast cancer

    * No concurrent chemotherapy for breast cancer
  * At least 1 month since prior and no concurrent treatment with corticosteroid
  * At least 2 weeks since prior and no concurrent use of antibiotics
  * At least 2 weeks
  * No history of chest wall irradiation
  * No presence of breast implants
  * No prior or concurrent tamoxifen within the past 90 days
  * No chronic/concurrent medications that inhibit platelet function, including any of the following:

    * Aspirin
    * Non-steroidal anti-inflammatory drugs (i.e., Aleve®, Motrin®, ibuprofen)
    * Coumadin
    * Heparin
    * Low molecular weight heparin
    * Anti-platelet agents

      * No prior short-term use of platelet inhibitors ≥ 7 days prior to RPFNA
  * No concurrent ingestion of the following:

    * Pumpkin seeds
    * Sesame seeds
    * Fish oil supplements
  * At least 30 days since prior and no concurrent flaxseed supplements, fish oil, or flaxseed oil
  * No concurrent treatment for another malignancy

Ages: 21 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2008-04; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Alteration in intermediate biomarkers of breast cancer risk at baseline and at 1, 3, and 6 months | 6 months

SECONDARY OUTCOMES:
Tolerability and compliance | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Swati Kulkarni, M.D., Principal Investigator — University of Chicago
Locations (2):
- United States (2):
  - University of Chicago Medicine, Chicago, Illinois
  - Roswell Cancer Park Institute, Buffalo, New York